CLINICAL TRIAL: NCT03322748
Title: Efficacy of Isometric Contraction Exercises of Lower Limbs Muscles, in Modulating Neurological Control of Bladder Function in Patients With Multiple Sclerosis
Brief Title: Efficacy of Lower Limb Exercises on Overactive Bladder Symptoms in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Giancarlo Comi, Director of Department of Neurology and Institute of Experimental Neurology, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OVERACT V1
Record Dates: First submitted 2017-10-13; First posted 2017-10-26 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Overactive Bladder Syndrome; Multiple Sclerosis; Muscle Strain
MeSH Terms: conditions — Multiple Sclerosis; Sprains and Strains

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Usual physical therapy+ strengthening of lower limbs muscles
  Interventions: Other: Usual physical therapy+ strengthening of lower limbs muscles
- Control group (Other): Usual physical therapy
  Interventions: Other: Usual physical therapy

INTERVENTIONS:
Other: Usual physical therapy+ strengthening of lower limbs muscles — Experimental group will perform usual physical therapy plus 3 series of isometric contractions of ankle plantarflexor and Hamstring muscles bilaterally, each lasting 5 seconds.
  Arms: Experimental group
Other: Usual physical therapy — Usual physical therapy
  Arms: Control group

SUMMARY:
The aim of the study (OVERACT_V1) is to verify if the isometric contraction of ankle plantarflexor and Hamstring muscles, induces a significant reduction of overactive bladder symptoms in patients with Multiple sclerosis.

DETAILED DESCRIPTION:
The aim of the study (OVERACT_V1) is to verify if the isometric contraction of ankle plantarflexor and Hamstring muscles, induces a significant reduction of overactive bladder symptoms in patients with Multiple sclerosis. It's known that the electric stimulation of the Posterior Tibial nerve induces an improvement of overactive bladder symptoms through a modulation of spinal circuitry, which occurs with unknown mechanisms. The investigators' hypothesis is that the voluntary muscular activation may induce a modulation of the sacral root as long as the electric stimulation. 30 patients will be recruited within 2 years, since October 2017 through October 2019. This is a monocentric, randomized controlled , in single blind, not pharmacological study.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis Patients
* Urge score >=2
* urinary daytime frequency >=8
* stable overactive bladder symptoms for 6 months
* MRC ( Medical Research Council) scale of ankle plantarflexors and hamstrings >=2
* signed informed consensus

Exclusion Criteria:

* FIM ( Functional Independence Measure) memory items <=4
* impairment in registering bladder diary
* inclusion in other experimental study
* specific straightening during the suty period
* PVR >= 200 ml ina single evaluation or PVR (post void residual) >=150 in 4 evaluation (twice a day for 2 consecutive days)
* Urinary infections
* concomitant urological disease
* intrathecal baclofen pump
* SANS (Stoller Afferent Nerve Stimulation)
* modification of therapy for overactive bladder symptoms within three months before entering the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change of Urinary frequency | at 6th and 22nd day
  mean of voluntary urination episodes daytime during 4 days of bladder diary
Change of Urge score | at 6th and 22nd day
  mean of score evaluating the perception of urge that patient experiences every urination. The subscale scores are:
  * 0, if patient doesn't need to urinate, but urinates before going out from home or concerned about the unavailability of toilet;
  * 1, if patient doesn't experience urgent urination;
  * 2, presence of urgency but disappeared before getting to the toilet;
  * 3, presence of urgency and reached the toilet without leakage of urine
  * 4, presence of urgency and did not reach the toilet with leakage of urine
Change of total score of OAB-q ( Overact Bladder questionnaire) long form | at 3rd and 18th day
  questionnaire evaluates the impact of overactive bladder symptoms on activities of daily living 8 ITEMS SYMPTOM BOTHER (each item has a subscale score from 1 to 6) + 25 ITEMS HEALTH-RELATED QUALITY OF LIFE (each item has a subscale score from 1 to 6)

SECONDARY OUTCOMES:
Change of Urine volume | at 6th and 22nd day
  Minimum , maximum and mean of urine volume voiding during 4 days of bladder diary
Change of episodes of urinary incontinence | at 6th and 22nd day
  Mean of involuntary leakage of urine during 4 days of bladder diary
Change of episodes of nocturia | at 6th and 22nd day
  Mean of voluntary urination episodes nightime during 4 days of bladder diary
Change of Postvoid Residual Volume | at 3rd and 18th day
  Mean of 3 measurement of Urine residual after voluntary voiding
Change of Pad-test 24 Hours | at 6th and 22nd day
  Mean of numbers and weight of pads
PGI (Patient global impression of improvement) | at 18th day
  Questionnaire on subjective impression of improvement of overactive bladder symptoms
Change of value at Uroflussimetry | at 3rd and 18th day
  Mean of maximum urinary flow rate (Qmax) value at uroflussimetry
Change of value at "H REFLEX" test | at 6th and 22nd day
  Evaluation of H wave mean amplitude and of Ratio of maximum H reflex to maximum M response after a train of stimuli given at 1 and 0.1 Hz
Change of EDSS (Expanded Disability Status Scale) | at 2nd and 22nd day
  Mean of value at EDSS that quantifying disability in multiple sclerosis
Change of Barthel Index Score | at 2nd and 22nd day
  Mean of total score measuring performance in activities of daily living
Change of MAS (Modified Ashworth Scale ) | at 2nd and 22nd day
  Mean of score (0-4) measuring spasticity of plantarflexors and Hamstring muscles

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Prof. Giancarlo Comi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No